CLINICAL TRIAL: NCT03356717
Title: Impact of the Use of an Observer Tool Based on Technical Skills on Learning Outcomes in Anesthesia Residents Undergoing High Fidelity Simulation
Brief Title: Effect of an Observer Tool on Learning Outcomes During High Fidelity Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Paris-Sud (Other)
Responsible Party: Principal Investigator, Dan Benhamou, Professor of Anesthesia and Intensive Care Medicine, Chair of the simulation center, Université Paris-Sud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UParis-Sud
Record Dates: First submitted 2017-06-22; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Simulation
Keywords: simulation, high-fidelity, observer tool; learning outcomes
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- educational intervention - observer tool (Experimental): Participants in this arm will be given the observer tool (OT) before the scenario and will be explained how to use it, i.e. observe all details of the scenario on the screen and tick on the OT all actions which are done by active participants.The observer tool will also be used to engage observers during the debriefing session.
  The scenario will then be observed in a screen (i.e. the scenario is played by active participants in an adjacent room using direct video-recording and transmission.
  Interventions: Behavioral: educational intervention with observer tool
- without observer tool (Active Comparator): Participants in this arm will not be given the observer tool (OT) before the scenario but will be asked to observe all details of the scenario on the screen.The observers will also be asked to participate during the debriefing session.
  Interventions: Behavioral: educational intervention

INTERVENTIONS:
Behavioral: educational intervention with observer tool — To assess if the use of an observer tool by observers during high fidelity simulation improves learning outcomes
  Arms: educational intervention - observer tool
Behavioral: educational intervention — without observer tool
  Arms: without observer tool

SUMMARY:
The increasing use of high-fidelity simulation is limited by the imbalance between the growing number of students and the human resources available in such a way that all residents cannot play a role during scenarios. The learning outcomes of observers need to be studied in more depth. Previous studies have provided controversial results but overall no significant differences in learning outcomes can be demonstrated between observers and participants engaged as players in scenarios.

Moreover, preliminary data suggest that learning outcomes of observers might be improved by using an observer tool during the scenario. However, no high-quality study has yet shown if this assumption is verified.

In the present study, 3rd-4th year residents in anesthesia will be randomized before high fidelity scenarios to act as observers only or active participants in some scenarios and observers in others.

The main outcome parameter will be the learning outcomes by comparing data obtained before and after the sessions by using questionnaires specifically dedicated to the knowledge of technical skills in the management of crisis scenarios.

DETAILED DESCRIPTION:
The increasing use of high-fidelity simulation in France during the anesthesia curriculum is limited by the imbalance between the growing number of students and the human resources available in such a way that all residents cannot play a role during scenarios. This leads to a new situation in which not all residents can be an active participant in scenarios with some remaining observers all along the simulation sessions. Based on Kolb experiential theory, this situation should lead to a decreased knowledge acquisition. Previous studies have however provided controversial results but overall no significant differences in learning outcomes can be demonstrated between observers and participants engaged as players in scenarios.

Moreover, preliminary data suggest that learning outcomes of observers might be improved by using an observer tool during the scenario. However, no high-quality study has yet shown if this assumption is verified.

In the present study, after informed consent will be obtained, 3rd-4th year residents in anesthesia will be randomized before high fidelity scenarios to act as observers only or active participants in some scenarios and observers in others.

The main outcome parameter will be the learning outcomes by comparing data obtained before and after the sessions by using questionnaires specifically dedicated to the knowledge of technical skills in the management of crisis scenarios. In addition, self-efficacy of the simulation sessions will be explored through the responses to additional questionnaires evaluating the change in non-technical skills after the sessions.

ELIGIBILITY:
Inclusion Criteria:

residents in anesthesia

Exclusion Criteria:

none

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Learning outcomes assessing knowledge of technical skills | measured before and immediately after the session
  The main outcome parameter will be the learning outcomes by comparing data obtained before and after the sessions by using questionnaires specifically dedicated to the knowledge of technical skills in the management of crisis scenarios: change will be assessed

SECONDARY OUTCOMES:
self assessment of the effect of the simulation session on non-technical skills | measured immediately after the session
  Self-efficacy of the simulation sessions will be explored through the responses to additional questionnaires evaluating the change in non-technical skills after the sessions

CONTACTS AND LOCATIONS:
Overall Officials: BENHAMOU Dan, MD, Principal Investigator — Université Paris-Sud
Locations (1):
- Université Paris Sud, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai A, Haligua A, Dylan Bould M, Everett T, Gale M, Pigford AA, Boet S. Learning crisis resource management: Practicing versus an observational role in simulation training - a randomized controlled trial. Anaesth Crit Care Pain Med. 2016 Aug;35(4):275-81. doi: 10.1016/j.accpm.2015.10.010. Epub 2016 Mar 14. PMID 26987738
- [Derived] Suet G, Blanie A, De Montblanc J, Benhamou D. Use of an Observer Tool to Enhance Observers' Learning of Anesthesia Residents During High-Fidelity Simulation: A Randomized Controlled Trial. Simul Healthc. 2022 Feb 1;17(1):e75-e82. doi: 10.1097/SIH.0000000000000584. PMID 34120134
- See also: Observer roles that optimise learning in healthcare simulation education: a systematic review. O'Regan et al. Advances in Simulation (2016) 1:4 — https://advancesinsimulation.biomedcentral.com/articles/10.1186/s41077-015-0004-8